CLINICAL TRIAL: NCT05042050
Title: Attachment-focused iMAgery Therapy for PSychosis (A-iMAPS): a Case Series
Brief Title: Attachment-focused iMAgery Therapy for PSychosis (A-iMAPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Pennine Care NHS Foundation Trust (Other Government); Greater Manchester Mental Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nicola Airey, Trainee Clinical Psychologist, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS001888
Record Dates: First submitted 2021-08-31; First posted 2021-09-13 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Psychosis; Psychosis-Related PTSD
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Proof of Concept Case Series Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-iMAPS Intervention (Experimental): Participants will receive six sessions of Attachment-focused iMAgery therapy for PSychosis. They will be randomised to different baseline lengths (two to five assessment sessions)
  Interventions: Behavioral: A-iMAPS

INTERVENTIONS:
Behavioral: A-iMAPS — Imagery therapy targeting Psychosis-Related PTSD

SUMMARY:
The relationships we have in childhood affect how we relate to others across our life, including how safe or secure we feel. If our caregivers do not meet our needs well enough in childhood, this can lead to an 'insecure attachment style'. This means we may push others away or cling to them, but never feel fully safe or secure with them. This style is common in people who have mental health problems. This includes psychosis, when people have unusual experiences such as hearing voices others cannot hear. A lot of people with psychosis have difficult experiences with mental health services. This includes involuntary treatments, traumatic interactions and hospital stays, where they may think staff are trying to harm rather than help them. As a result they may not feel safe working with staff and they might re-experience the negative memories of these events. This is known as psychosis-related Post-Traumatic Stress Disorder (PR-PTSD) and can lead to ongoing problems.

Imagery is often defined as mental pictures but it includes imagining our senses (smell, touch, taste) too. It can be a useful therapy tool to help people to work with difficult memories and can help them to feel more safe and secure. Research shows that this is helpful for people with psychosis and people who have been through trauma. Hence, it may be helpful for people with PR-PTSD. The study aims to see if it is viable to do a 6-session therapy using imagery to target PR-PTSD memories. The study will use a case series design where up to 12 people with psychosis will be able to try the therapy. They will be asked to complete questionnaires to understand any potential benefits of the therapy. The findings could inform the research and allow for further development of therapies in this area.

DETAILED DESCRIPTION:
Attachment theory underpins human interpersonal experience: it suggests that our early relationships, typically those with our primary caregivers in infancy, have a profound effect on how we learn to relate to the others across the lifespan. Attachment styles in adulthood, particularly insecure styles, have been associated with mental health problems, and it has been noted that improving attachment security can improve mental health.

In the last decade, there has been an increase in research around the role of attachment in psychosis, with an over-representation of insecure attachment patterns seen in individuals with such diagnoses (76% in psychosis compared to 38% in non-clinical samples). A number of studies have identified links with insecure attachment in several aspects of psychopathology, including voice-hearing, persecutory delusions, social functioning and negative symptoms, though the mechanisms between such remain poorly understood.

Attachment insecurity is significantly associated with paranoia and recent research has focused on reducing this using the concept of "felt security", which is defined as "a sense of interpersonal safety associated with secure, protective relationships". In childhood, this sense of safety and security constitutes a 'secure base' from which the child is able to explore. Priming felt security through imagery (i.e. undertaking an imagery exercise focused on secure attachment with another individual in the image) has been found to reduce paranoia in non-clinical adult samples. Moreover, 'felt security' imagery has been deemed effective in engendering a sense of security and reducing paranoia prior to rescripting trauma memories with an individual with psychosis.

Imagery interventions have been long established for use as part of therapy for individuals with psychosis, and have been recognised as a frontier in therapeutic intervention across disorders, including working with negative imagery (e.g., imagery rescripting) and positive imagery. A case series was completed and subsequently a protocol published for a six-session imagery intervention, iMAgery focused psychological therapy for persecutory delusions in PSychosis (iMAPS), targeting intrusive mental imagery and negative beliefs about self and others in psychosis with a combination of negative and positive imagery techniques, which indicated feasibility of combining various imagery techniques in a short intervention for psychosis.

Individuals with psychosis may not only experience intrusive images as a component of their psychotic symptomology, but also as a consequence of their psychosis itself. Psychosis-Related Post-Traumatic Stress Disorder (PR-PTSD) is an under-researched area but a recent review suggested that between 14% and 47% of individuals with psychosis may have PR-PTSD, with associated factors including symptomology of psychosis, treatment factors (involuntary admissions, traumatic inpatient events, restraint) and attachment style. However, there appears to be minimal published literature on this beyond first-episode psychosis. Anxiety in attachment relationships has been identified as positively correlated with psychosis-related and hospital-related PTSD symptoms.

The present study aims to add to the limited literature on PR-PTSD by evaluating the feasibility of a short six-session attachment-focused imagery intervention for psychosis, based upon the iMAPS protocol, which will be adapted to include 'felt security' imagery and the imagery rescripting will focus on psychosis-related trauma. It is anticipated that this would reduce PTSD symptomology. Moreover, by using attachment security primes in conjunction with rescripting, paranoia may also be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Is currently receiving care under an NHS Community Mental Health Team, and meets ICD-10 or ICD-11 criteria for a schizophrenia-spectrum diagnosis (schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder or psychotic disorder not otherwise specified) indicated by case notes, or under the care of an Early Intervention in Psychosis Service
* Aged 16 or above
* Medication stable for ≥ one month, as indicated by their Care Coordinator
* Has capacity to give written, informed consent
* Proficient in English to complete study questionnaires
* A score of one or more on the four psychosis-related trauma items (items 15 to 18) on the Trauma and Life Events Checklist (Carr et al., 2018b)

Exclusion Criteria:

* Has an acquired brain injury
* Has a history of substance misuse that is judged to be the acute cause of the psychotic experiences
* Currently experiencing an acute episode requiring inpatient care
* Currently undertaking psychological therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Number of participants approached and recruited to the intervention | Throughout recruitment phase of the study, an average of 24 weeks
Number of sessions attended | Throughout the study, attendance recorded for each intervention session, an average of 1 year
  Calculated as a percentage
Number of participants who drop out of the intervention | For the duration of the study, an average of 1 year
  Including the point at which they drop out
Number of Adverse Events and Serious Adverts Events recorded during the study | For the duration of the study, an average of 1 year

SECONDARY OUTCOMES:
The suitability of outcome measures used, determined by the number completed | For the duration of the study, an average of 1 year
  Calculated as a percentage, outcome measures completed weekly
Change from baseline in PTSD score | For duration of intervention, up to 12 weeks
  Measured by the PTSD checklist for DSM-5, scored 0 to 80, higher score suggesting worsening symptoms. Once a week from baseline to end of therapy assessment
Change from baseline in paranoia score | For duration of intervention, up to 12 weeks
  Measured using the Revised Green Paranoid Thoughts Scale, scored 0 to 40, higher score suggests worsening symptomology. Once at initial baseline appointment and once at end of therapy assessment
Change from baseline in core schemas | For duration of intervention, up to 12 weeks
  Measured using the Brief Core Schema Scale, scored 0 to 24 on four scales (positive-self, negative-self, positive-others, negative-others), higher score on positive scales suggests improvements, higher score on negative scales suggests worsening. Once at initial baseline appointment and once at end of therapy assessment
Change from baseline in attachment style | For duration of intervention, up to 12 weeks
  Measured using the Revised Psychosis Attachment Measure to determine if style changes. Once at initial baseline appointment and once at end of therapy assessment
Change from baseline in felt security | For duration of intervention, up to 12 weeks
  Measured using an adapted version of the Felt Security Scale, scored 6 to 36, higher score indicates higher levels of felt security. Weekly at each baseline assessment, twice in each therapy session (pre and post attachment prime), and one final at end of therapy assessment

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Berry, PhD, Principal Investigator — University of Manchester
Locations (1):
- Pennine Care NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated anonymised participant data

REFERENCES:
- [Background] Mikulincer M, Shaver PR. An attachment perspective on psychopathology. World Psychiatry. 2012 Feb;11(1):11-5. doi: 10.1016/j.wpsyc.2012.01.003. PMID 22294997
- [Background] Carr SC, Hardy A, Fornells-Ambrojo M. Relationship between attachment style and symptom severity across the psychosis spectrum: A meta-analysis. Clin Psychol Rev. 2018 Feb;59:145-158. doi: 10.1016/j.cpr.2017.12.001. Epub 2017 Dec 6. PMID 29229220
- [Background] Lavin R, Bucci S, Varese F, Berry K. The relationship between insecure attachment and paranoia in psychosis: A systematic literature review. Br J Clin Psychol. 2020 Mar;59(1):39-65. doi: 10.1111/bjc.12231. Epub 2019 Aug 7. PMID 31390076
- [Background] Bullock G, Newman-Taylor K, Stopa L. The role of mental imagery in non-clinical paranoia. J Behav Ther Exp Psychiatry. 2016 Mar;50:264-8. doi: 10.1016/j.jbtep.2015.10.002. Epub 2015 Oct 8. PMID 26492591
- [Background] Pitfield C, Maguire T, Newman-Taylor K. Impact of attachment imagery on paranoia and mood: evidence from two single case studies. Behav Cogn Psychother. 2020 Sep;48(5):572-583. doi: 10.1017/S1352465820000351. Epub 2020 Jun 29. PMID 32594948
- [Background] Morrison AP. The use of imagery in cognitive therapy for psychosis: a case example. Memory. 2004 Jul;12(4):517-24. doi: 10.1080/09658210444000142. PMID 15487547
- [Background] Holmes EA, Mathews A, Dalgleish T, Mackintosh B. Positive interpretation training: effects of mental imagery versus verbal training on positive mood. Behav Ther. 2006 Sep;37(3):237-47. doi: 10.1016/j.beth.2006.02.002. Epub 2006 May 24. PMID 16942975
- [Background] Taylor CDJ, Bee PE, Kelly J, Emsley R, Haddock G. iMAgery focused psychological therapy for persecutory delusions in PSychosis (iMAPS): a multiple baseline experimental case series. Behav Cogn Psychother. 2020 Sep;48(5):530-545. doi: 10.1017/S1352465820000168. Epub 2020 Apr 8. PMID 32264985
- [Background] Buswell G, Haime Z, Lloyd-Evans B, Billings J. A systematic review of PTSD to the experience of psychosis: prevalence and associated factors. BMC Psychiatry. 2021 Jan 7;21(1):9. doi: 10.1186/s12888-020-02999-x. PMID 33413179